CLINICAL TRIAL: NCT02068053
Title: Pharmacokinetics and Metabolism of [14C] BMS-986020 in Healthy Male Subjects
Brief Title: Absorption, Distribution, Metabolism and Excretion (ADME) Study of BMS-986020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IM136-006
Record Dates: First submitted 2014-02-19; First posted 2014-02-20 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Immunosuppression For Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A - BMS-986020 (Experimental): 600 mg (approximately 80 micro Curie) of [14C] BMS-986020 Single Dose for 1 Day (Day 1) orally
  Interventions: Drug: [14C] BMS-986020

INTERVENTIONS:
Drug: [14C] BMS-986020
  Other Names: Lysophosphatidic Acid receptor 1 (LPA1) Antagonist

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), metabolism, routes and extent of elimination, as well as safety and tolerability of a single oral solution dose of [14C] Bristol-Myers Squibb (BMS)-986020 in healthy male subjects.

DETAILED DESCRIPTION:
Primary purpose: Other - This study will investigate the pharmacokinetic, biotransformation, routes of elimination, and mass balance of BMS-986020 in humans. The knowledge of the routes of elimination of the drug and its metabolites is useful for evaluating the likelihood of effects of renal or hepatic impairment on the disposition of BMS-986020

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy male subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Body weight of at least 50 kg (110 lbs), Body mass index (BMI) of 18.0 to 32.0 kg/m2, inclusive. Body mass index = weight (kg)/[height(m)]2
* Men, ages 18 to 50 years, inclusive
* Men who are sexually active with women of childbearing potential (WOCBP) (except those with vasectomy with documented azoospermia 90 days after procedure) must agree to follow instructions for method(s) of contraception for the duration of treatment plus 5 half-lives of the investigational drug (4 days) plus 90 days (duration of sperm turnover) for a total of 94 days post-treatment completion

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Current or recent history of constipation or irregular bowel movements (less than once per 2 days)
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery that could impact upon the absorption of study drug, including cholecystectomy
* History of Gilbert's Syndrome
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma only)
* Blood transfusion within 4 weeks of study drug administration
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access
* Recent (within 6 months of study drug administration) history of smoking
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations beyond what is consistent with the target population
* History of allergy to LPA1 antagonists or related compounds

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986020 and Total Radioactivity (TRA) | 22 Timepoints up to Day 11
Time of maximum observed plasma concentration (Tmax) of BMS-986020 and TRA | 22 Timepoints up to Day 11
Area under the concentration time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) of BMS-986020 and TRA | 22 Timepoints up to Day 11
Area under the concentration time curve from time zero to 168 hours postdose (AUC(0-168)) of BMS-986020 and TRA | 19 Timepoints up to Day 8
Area under the concentration time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-986020 and TRA | 22 Timepoints up to Day 11
Terminal plasma half-life (T-Half) of BMS-986020 and TRA | 22 Timepoints up to Day 11
Apparent total body clearance (CL/F) of BMS-986020 | 19 Timepoints up to Day 8
Percent of plasma BMS-986020 AUC(0-T) (%AUC(0-T)) relative to plasma TRA AUC(0-T) | 22 Timepoints up to Day 11
Percent of plasma BMS-986020 AUC(INF) (%AUC(INF)) relative to plasma TRA AUC(INF) | 22 Timepoints up to Day 11
Percent of total administered radioactivity excreted in urine (% UR) | 13 Timepoints up to Day 11
Percent of total administered radioactivity excreted in feces (% FE) | 11 Timepoints up to Day 11
Percent of total administered radioactivity recovered in urine and feces (%TOTAL) | 13 Timepoints up to Day 11

SECONDARY OUTCOMES:
Incidence of Adverse Event (AE)s collected during the study will be reviewed for potential significance and clinical importance | Upto Day 11
Clinical laboratory test results: Safety laboratory testing will be drawn at specified times | Up to Day 11
Vital Signs: Blood pressure, heart rate, respiratory rate, and body temperature measurements will be assessed at specified time points | Up to Day 11
Electrocardiogram (ECG): Regular ECG endpoints (heart rate, PR interval, QRS interval, and QT intervals corrected for heart rate) and investigator identified abnormalities will be assessed at the time points | Up to Day 11
Physical examinations: Physical examinations will be assessed at the time points | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb